CLINICAL TRIAL: NCT06517797
Title: Phase IIb Placebo-Controlled Double-Blind Randomized Parallel Groups Study to Determine the Efficacy and Safety of S1B-509 for Weight Loss
Brief Title: One-Year Study of S1B-509 vs Placebo for Weight Loss
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: S1 Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S1B-509-2000
Record Dates: First submitted 2024-07-15; First posted 2024-07-24 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: S1B-509; diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Parallel assignment to putatively active treatment at low and high dose or placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: tablets of one of the actives and capsules of the other active matched to placebo tablets and capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- S1B-509 (proprietary combination of trazodone and bupropion) low dose (Experimental): Simultaneous oral dosing once daily with two to four extended-release tablets or capsules of S1B-509, for 48 weeks
  Interventions: Drug: S1B-509 low dose
- Placebo (Placebo Comparator): Simultaneous oral dosing once daily with two to four placebos, for 48 weeks
  Interventions: Drug: Placebo
- S1B-509 (proprietary combination of trazodone and bupropion) high dose (Experimental): twice the dose of "S1B-509 low dose"
  Interventions: Drug: S1B-509 High Dose

INTERVENTIONS:
Drug: S1B-509 low dose — S1B-509 has multiple neurotransmitter activities
  Other Names: proprietary combination of trazodone and bupropion at low dose
  Arms: S1B-509 (proprietary combination of trazodone and bupropion) low dose
Drug: Placebo — matched pills to S1B-509
  Arms: Placebo
Drug: S1B-509 High Dose — S1B-509 has multiple neurotransmitter activities
  Other Names: proprietary combination of trazodone and bupropion at high dose
  Arms: S1B-509 (proprietary combination of trazodone and bupropion) high dose

SUMMARY:
This is a study to test whether S1B-509 given orally daily helps people with overweight or obesity to lose more weight than with placebo over a year.

DETAILED DESCRIPTION:
This trial is to determine proof of concept for S1B-509 vs. placebo and to define a suitable dose escalation scheme and range for S1B-509 regarding safety, tolerability, and efficacy. The treatments will be given along with dietary advice and food intake monitoring. Change in body weight and in measures relating to obesity and its complications such as diabetes will be measured from baseline to week 48. Safety will be determined from adverse event reports, vital signs, routine laboratory tests, and mental health screeners.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obesity disease and inadequately controlled body weight with diet and/or exercise
* Body mass index (BMI) ≥ 27 kg/m2 with significant comorbidity, e.g., type 2 diabetes, hypertension, dyslipidemia, sleep apnea, cardiovascular disease
* Waist circumference at umbilical level ≥ 85 cm for male, ≥ 90 cm for female
* Visceral fat area ≥ 100 cm2
* Agreement to comply with the study-required life-style intervention and treatment during the full duration of the study.
* Side effects from any continuing concomitant medications must be mild and stable or nil.
* Females: not pregnant or lactating for six months; using medically reliable contraception, i.e., diaphragm or (male or female) condom and spermicide, IUD, tubal sterilization, hormonal contraception (oral, vaginal, or implant), or (if the investigator finds the patient credibly monogamous) vasectomy of male partner.
* Gives informed consent for and is willing to undergo all of the scheduled evaluations.
* Prompt for screening and baseline visits, is cooperative, and takes reasonable directions without excessive explanations.

Exclusion Criteria:

1. Use of pharmacologically active weight-loss medications, glucagon-like peptide-1 (GLP-1) agonists or sodium-glucose co-transporter 2 (SGLT2) inhibitors, within 3 months of screening, or between screening and randomization.
2. Use of alpha glucosidase inhibitors within 3 months of Visit 1, or between screening and randomization.
3. Bariatric surgery
4. Lack of compliance with lifestyle intervention (defined as weight gain during 4-week Screening/run-in or with study medication (defined as < 80% study drug intake in more than one 4-week period
5. History of ketoacidosis, lactic acidosis, or hyperosmolar coma, or any of these occurring between Visit 1 and 2/randomization
6. Diabetics with HbA1c levels over 10 percent or fasting glucose levels greater than or equal to 270 mg/dl.
7. Symptomatic infection in the 4 weeks prior to screening or randomization.
8. Gastro-intestinal (GI) disorders associated with chronic diarrhea.
9. Congestive heart failure, New York Heart Association (NYHA) class III or IV
10. Body dysmorphic disorder or compulsive eating disorder
11. Chronic conditions that may in the investigator's judgment be expected to be unstable and affect overall health are not allowed. Examples: gastrointestinal bleeding in prior 6 months, diabetes mellitus with HB A1C >8.9, asthma not well controlled with treatment once or twice daily, current Major Depressive Disorder or recurrence of MDD off treatment for at least 2 months, anxiety disorder severe enough to prevent employment, severe sleep apnea, history within the prior year of suicidality or drug abuse, history of active breast, cervical, uterine, ovarian or other systemic cancer within the prior 24 months.
12. Requires CYP3A4, CYP 2B6, or CYP 2D6 strong inhibitor or inducer drugs
13. Takes any sex hormone other than an approved hormonal contraceptive
14. Takes an antiepileptic/mood stabilizer, antipsychotic, antidepressant, anxiolytic, or hypnotic drug
15. Drinks more than 7 alcoholic drinks per week (12-oz beer, 4-oz wine, 1 ½ oz liquor etc)
16. Uses marijuana more than once a week
17. History of seizures as an adult or use of antiepileptic medication
18. Long QT syndrome (QTc <=480 msec), other significant cardiovascular disease (hypertension controlled with one medication is acceptable)
19. Moderate or severe dysfunction of the liver (any LFT >=3x ULN) or renal dysfunction (BUN > 30 or Cr >2.0)
20. Uses sedating antihistamines or prescription sedatives daily
21. History of blood clots or abnormal bleeding tendencies, including daily use of medications adversely affecting coagulation, e.g., NSAIDs, systemic corticosteroids, or >81 mg aspirin daily.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Per cent weight change | 48 weeks
  100 (Weight at follow-up) - (weight at baseline)/(weight at baseline)
Proportion losing at least 5% body weight | 48 weeks
  (number of subjects (no. ss) per group losing at least 5% body weight)/(total no. ss/group

SECONDARY OUTCOMES:
Waist circumference | 48 weeks
  measured waist in inches or centimeters
Proportion losing 10% | 48 weeks
  per cent of patients per group losing ten percent weight, a substantial amount
Proportion losing 15% | 48 weeks
  per cent of patients per group losing a highly substantial amount of weight
Change in systolic blood pressure | 48 weeks
  average gain in systolic blood pressure per group
Change in diastolic blood pressure | 48 weeks
  average change in diastolic pressure per group
Change in Hemoglobin A1c | 48 weeks
  change in glycosylated hemoglobin, a measure of diabetes; normal is less than 6.5%
Change in Columbia suicidality screener | 48 weeks
  6 yes/no items, patient-rated screener on suicide ideation and behavior, "no" on each is best
Change in Personal Health Questionnaire, 9-item version | 48 weeks
  depression screener. Sum of 9 self-rated items from 0 (best) to 3 (worst).
Adverse events | 4 weeks
  Change in subjective (answer to "how have you felt" or objective findings
Change in Female Sexual Function Index, Female | 4 weeks
  19-item self-rated scale on sexual response, sum of ratings from 0 or 1 (worst) to 5 (best)
Change in International Index of Erectile Function, 5-item version | 4 weeks
  5-item self-rated scale on erectile function, sum of items rated from 1 (worst) to 5 (best)
Edmonton Obesity Staging System | 4 weeks
  Single-item categorical rating from 0 (normal) to 4 (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas E Sitchon, B.S., Study Chair — S1 Biopharma, Inc.

IPD SHARING:
Plan to Share IPD: No